CLINICAL TRIAL: NCT00192049
Title: A Randomized Phase II Study Comparing Single Agent Gemcitabine Intravesical Therapy Versus Mitomycin C in Patients With Intermediate Risk Superficial Bladder Cancer
Brief Title: A Randomized Study Comparing Single Agent Gemcitabine Intravesical Therapy Versus Mitomycin C in Patients With Intermediate Risk Superficial Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8048; B9E-MC-S344
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Superficial Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine; Mitomycin

INTERVENTIONS:
Drug: Gemcitabine
Drug: mitomycin C

SUMMARY:
Gemcitabine has been shown to be highly effective and well tolerated in the first and second line therapy, as a single agent or in combination therapy for treatment of metastatic transitional cell carcinoma. On the basis of Gemcitabine clinical activity and good tolerability this drug has been recently tested in intravesical therapy. we consider Gemcitabine as a good therapy candidate for patient with intermediate risk superficial bladder cancer. Based on the phase I/II clinical trials w are going to explore the efficacy and tolerability of Gemcitabine in this setting, and compare it to Mitomycin C which is widely used in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified superficial transitional cell carcinoma of the bladder.
* patients with primary or recurrent intermediate risk superficial bladder cancer after TUR. Patients with primary tumor with stage TaG1 with multiple lesions (>3) or lesions bigger than 3 cm or patients with TaG2-3 or T1G1-2.
* Patients must not be pre-treated with any intravesical immunotherapy (BCG) or chemotherapy.
* Male or female, age greater than 18.

Exclusion Criteria:

* Time between TUR and start of intravesical chemotherapy will be longer than 4 weeks.
* Patients who have received previous (BCG) or chemotherapy.
* Patients with evidence of invasive, locally advanced or metastatic bladder cancer (greater than or equal to T2 disease; stage greater than or equal to B1) or patients with upper urinary tract disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2003-12; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Compare the tumor recurrence rate at 12 months after TUR in patients with intermediate risk superficial bladder cancer treated with intravesical Gemcitabine or Mitomycin C.

SECONDARY OUTCOMES:
Tumor recurrence rate in 6 months
disease free interval
Toxicity profile (local and systemic)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon -Fri 9 AM-5 PM Eastern time (UTC/GMT - 5 hours,EST), Study Director — Eli Lilly and Company
Locations (5):
- Israel (5):
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Beersheba
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Haifa
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Jerusalem
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Kfar Saba
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Tel Litwinsky

REFERENCES:
- [Derived] Han MA, Maisch P, Jung JH, Hwang JE, Narayan V, Cleves A, Hwang EC, Dahm P. Intravesical gemcitabine for non-muscle invasive bladder cancer. Cochrane Database Syst Rev. 2021 Jun 14;6(6):CD009294. doi: 10.1002/14651858.CD009294.pub3. PMID 34125951
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com